CLINICAL TRIAL: NCT01372748
Title: Trial Of Continuous Compressions Versus Standard CPR In Patients With Out-Of-Hospital Cardiac Arrest
Brief Title: Continuous Chest Compressions vs AHA Standard CPR of 30:2
Acronym: CCC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Canadian Institutes of Health Research (CIHR) (Other Government); Heart and Stroke Foundation of Canada (Other); American Heart Association (Other); Defence Research and Development Canada (Industry); U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Principal Investigator, Susanne May, Principal Investigator, University of Washington
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 40404-B; 5U01HL077863-07 (NIH)
Record Dates: First submitted 2011-06-02; First posted 2011-06-14 (Estimated); Results first posted 2016-10-05 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2016-11

CONDITIONS: Out of Hospital Cardiac Arrest
Keywords: cardiac arrest; cardiopulmonary resuscitation
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard CPR (Active Comparator): American Heart Association (AHA)recommended cardiopulmonary resuscitation (CPR) of 30 compressions with brief pause for 2 ventilations
  Interventions: Other: Standard CPR
- Continuous chest compressions (Experimental): Continuous compression CPR
  Interventions: Other: Continuous chest compressions

INTERVENTIONS:
Other: Standard CPR — 30:2 CPR consists of 3 cycles of standard CPR with each cycle consisting of 30 chest compressions with a pause for 2 ventilations at a compression:ventilation ratio of 30:2. CCC consists of a series of three cycles of continuous chest compressions without pauses for ventilation. In either group, each cycle will be followed by rhythm analysis until three cycles are completed or restoration of spontaneous circulation (ROSC), whichever occurs first.
  Arms: Standard CPR
Other: Continuous chest compressions — Continuous chest compressions during the first 6 minutes of the resuscitation.
  Arms: Continuous chest compressions

SUMMARY:
The primary aim of the trial is to compare survival to hospital discharge after continuous chest compressions (CCC) versus standard American Heart Association (AHA) recommended cardiopulmonary resuscitation (CPR) with interrupted chest compressions (ICC) in patients with out-of-hospital cardiac arrest (OOHCA). The primary null hypothesis will be that the rate of survival to hospital discharge is not affected by use of continuous compressions with passive or positive pressure ventilation (intervention group) versus CPR with compressions interrupted for ventilation at a ratio of 30:2 (control group).

DETAILED DESCRIPTION:
The primary aim of the trial is to compare survival to hospital discharge after continuous chest compressions (CCC) versus standard American Heart Association (AHA) recommended cardiopulmonary resuscitation (CPR) with interrupted chest compressions (ICC) in patients with out-of-hospital cardiac arrest (OOHCA). For this study, CCC consists of a series of three cycles of continuous chest compressions without pauses for ventilation followed by rhythm analysis or until restoration of spontaneous circulation (ROSC), whichever occurs first. ICC consists of series of three cycles of standard CPR each cycle comprised of chest compressions with interposed ventilations at a compression:ventilation ratio of 30:2 (per AHA guidelines) followed by rhythm analysis or until ROSC, whichever occurs first. In either patient group, the duration of manual CPR before the first rhythm analysis will be 30 seconds or 120 seconds. This treatment period will be followed by two cycles of compressions then rhythm analysis (i.e. each of approximately 2 minutes duration) in either group. Other aims of the trial are to compare survival to discharge among patients grouped by first-recorded rhythm or other a priori subgroups, as well as to compare neurological status at discharge, mechanistic outcomes or adverse events between control and intervention groups.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or more (or local age of consent);
* Initial fire/Emergency Medical Services (EMS) chest compressions provided by Resuscitation Outcomes Consortium (ROC) study participating agency dispatched to the scene;
* Lack of the exclusion criteria below

Exclusion Criteria:

* EMS witnessed arrest;
* Written do not attempt resuscitation (DNAR) orders;
* Obvious primary asphyxia or respiratory cause of arrest (drowning, strangulation, hanging)
* Advanced airway placed prior to ROC EMS arrival, or pre-existing tracheostomy
* Traumatic cause (blunt, penetrating, burn) of arrest;
* Known prisoners;
* Known pregnancy;
* Uncontrolled bleeding or exsanguination
* Mechanical compression device used during study-assigned compression cycles

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23711 (Actual)
Dates: Start 2011-06; Primary Completion 2015-08 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Myron Weisfeldt, MD, MD, Study Chair — Johns Hopkins University
Locations (7):
- United States (5):
  - Alabama Resuscitation Center, Birmingham, Alabama
  - The Pittsburgh Resuscitation Network, University of Pittsburgh, Pittsburgh, Pennsylvania
  - Dallas Center for Resuscitation Research, University of Texas Southwestern Medical Center, Dallas, Texas
  - Seattle-King County Center for Resuscitation Research, Seattle, Washington
  - Milwaukee Resuscitation Network, Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (2):
  - University of Ottawa/University of British Columbia Collaborative RCC, Ottawa Health Research, Ottawa, Ontario
  - Rescu, Toronto, Ontario

REFERENCES:
- [Derived] Nichol G, Leroux B, Wang H, Callaway CW, Sopko G, Weisfeldt M, Stiell I, Morrison LJ, Aufderheide TP, Cheskes S, Christenson J, Kudenchuk P, Vaillancourt C, Rea TD, Idris AH, Colella R, Isaacs M, Straight R, Stephens S, Richardson J, Condle J, Schmicker RH, Egan D, May S, Ornato JP; ROC Investigators. Trial of Continuous or Interrupted Chest Compressions during CPR. N Engl J Med. 2015 Dec 3;373(23):2203-14. doi: 10.1056/NEJMoa1509139. Epub 2015 Nov 9. PMID 26550795
- [Derived] Brown SP, Wang H, Aufderheide TP, Vaillancourt C, Schmicker RH, Cheskes S, Straight R, Kudenchuk P, Morrison L, Colella MR, Condle J, Gamez G, Hostler D, Kayea T, Ragsdale S, Stephens S, Nichol G; ROC Investigators. A randomized trial of continuous versus interrupted chest compressions in out-of-hospital cardiac arrest: rationale for and design of the Resuscitation Outcomes Consortium Continuous Chest Compressions Trial. Am Heart J. 2015 Mar;169(3):334-341.e5. doi: 10.1016/j.ahj.2014.11.011. Epub 2014 Nov 20. PMID 25728722

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In this cluster randomized crossover trial, there are situations where age and gender are not known prior to the treatment being administered. These missing data account for the discrepancy between the enrollment number in the protocol section (23,711) and those in the participant flow module (23,687).
Period: Overall Study
Arm/Group | Standard CPR | Continuous Chest Compressions
Started | 11045 | 12642
Completed | 11022 (defined as having vital status) | 12603 (defined as having vital status)
Not Completed | 23 | 39
Not completed — Lost to Follow-up | 16 | 34
Not completed — Withdrawal by Subject | 7 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard CPR | Continuous Chest Compressions | Total
Number analyzed (Participants) | 11045 | 12642 | 23687
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (17.0) | 66.4 (17.2) | 66.3 (17.1)
Gender [Count of Participants; unit: Participants]
  Female | 3926 | 4618 | 8544
  Male | 7119 | 8024 | 15143
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 14 | 12 | 26
  Asian | 123 | 140 | 263
  Native Hawaiian or Other Pacific Islander | 23 | 28 | 51
  Black or African American | 1246 | 1350 | 2596
  White | 1795 | 1931 | 3726
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 7841 | 9180 | 17021
Region of Enrollment [Number; unit: participants]
  Canada | 6711 | 8010 | 14721
  United States | 4334 | 4632 | 8966

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Survive From the Time of Cardiac Arrest to Hospital Discharge
Description: Patients may die in the field (outside of the hospital at the time of the cardiac arrest), at the emergency room, in the hospital, or they are discharged alive from the hospital.
Time Frame: Patients will be followed from the time of the cardiac arrest until death or hospital discharge, whichever occurs first.
Population: The primary aim of the trial is to compare survival to hospital discharge after continuous chest compressions (CCC) versus standard American Heart Association (AHA) recommended cardiopulmonary resuscitation (CPR) with interrupted chest compressions (ICC) in patients with out-of-hospital cardiac arrest (OOHCA).
Measure: Number; unit: participants
Arm/Group | Standard CPR | Continuous Chest Compressions
Number analyzed (Participants) | 11022 | 12603
participants | 1072 | 1127

2. Secondary Outcome: Percentage of Participants Scoring at or Below a 3 on the MRS Scale
Description: Neurologic status at discharge will be assessed using the modified Rankin Score (MRS). A higher value indicates a worse outcome. 0-No symptoms at all; 1-No significant disability despite symptoms; able to carry out all usual duties and activities, 2-Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance, 3-Moderate disability; requiring some help, but able to walk without assistance; 4-Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance, 5-Severe disability; bedridden, incontinent and requiring constant nursing care and attention; 6-Dead
Time Frame: Patients will be followed from the time of the cardiac arrest until death or hospital discharge, whichever occurs first.
Measure: Number; unit: percentage of participants
Arm/Group | Standard CPR | Continuous Chest Compressions
Number analyzed (Participants) | 10892 | 12550
percentage of participants | 7.7 | 7.0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time a participating agency arrived on scene and up to 24 hours after Emergency Department arrival
Description: The following are commonly observed in patients who experience cardiac arrest or resuscitative efforts, and may or may not be attributable to specific resuscitation therapies. These were monitored and reported but not considered as adverse events of the study intervention. These include, but not limited to: pulmonary edema, airway bleeding, death, Clinical diagnoses of pneumonia, sepsis, cerebral bleeding, stroke, seizures, rearrest, serious rib fractures, and sternal fractures.
Arm/Group | Standard CPR | Continuous Chest Compressions
Serious Adverse Events (participants affected / at risk) | 0/11045 | 0/12642
Other Adverse Events (participants affected / at risk) | 1197/11045 | 1310/12642
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Standard CPR (N=11045) | Continuous Chest Compressions (N=12642)
Airway Bleed (Respiratory, thoracic and mediastinal disorders) | 764 | 881
Emesis (Gastrointestinal disorders) | 1197 | 1310
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1072 | 1137

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less